CLINICAL TRIAL: NCT04937491
Title: Detection of Minor Changes in Fluid Volume or Tonicity in Healthy Volunteers.
Acronym: CTR025
Status: Suspended | Type: Observational
Why Stopped: Due to covid-19
Sponsor: Mode Sensors AS (Industry)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: CTR025 HYDRA TROMSØ
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Healthy Nutrition
Keywords: dehyration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum: sodium, albumin, carbamide, glucose, creatinine and haemoglobin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Adult healthy volunteers (students). Intervention 1: Intake of water (2% of body weight) Intervention 2: Intake of sports drink (2% of body weight) Intervention 3: Intake of soya saus (salt): 10 ml (equal to 8 g salt) Intervention 4: Intake of 90 g sugar (jelly figures)
  Interventions: Device: New medical device (ReBalans)

INTERVENTIONS:
Device: New medical device (ReBalans) — Body worn, battery powered bioimpedance measuring patch device.

SUMMARY:
This study is aimed at detecting minor changes in hydration volume and tonicity. We will use healthy students of both sexes who will ingest fluids and nutrition that should lead to specific changes in both intracellular and extracellular volumes. The protocol is based on laboratory exercises previously carried out at The Arctic University of Norway (UiT).

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteer

Exclusion Criteria:

* Kidney disease,
* neurological,
* heart or endocrine disease,
* hypertension.
* Eating disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy volunteers (students), 20 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Ability to detect tonicity or volume change | 1 week
  Accurately depict each of the four interventions with a sensitivity better than 0.9.

CONTACTS AND LOCATIONS:
Locations (1):
- Arctic University of Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.